CLINICAL TRIAL: NCT03675633
Title: Fractional Excretion of Urea: an Excellent Simple Tool for the Differential Diagnosis of Acute Kidney Injury in Liver Cirrhosis
Brief Title: Fractional Excretion of Urea for the Differential Diagnosis of Acute Kidney Injury in Liver Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nermeen mahmoud mobarez, Doctor, Assiut University
Other Study IDs: FEUrea in liver cirrhosis
Record Dates: First submitted 2018-09-15; First posted 2018-09-18 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FEUrea in decompensated liver cirrhosis: FEUrea for the differential diagnosis of AKI in patients with cirrhosis and ascites Specifically, the ability of FEUrea to distinguish between ATN versus Pre renal azotemia and HRS
  Interventions: Diagnostic Test: FEUrea

INTERVENTIONS:
Diagnostic Test: FEUrea — FEUrea in decompansated liver cirrhosis

SUMMARY:
The aim of this study is to evaluate the diagnostic performance of FEUrea for the differential diagnosis of AKI in patients with cirrhosis and ascites Specifically, the ability of FEUrea to distinguish between ATN versus Pre renal azotemia and HRS.

DETAILED DESCRIPTION:
AKI according to KDIGO guidelines is defined as the followings:

* An increase in serum creatinine by ≥0.3 mg/dl (≥26.5 µmol/l) within 48 h
* An increase in serum creatinine to ≥1.5 times baseline within the previous 7 days
* Urine volume ≤0.5 ml/kg/h for 6 h Serum creatinine overestimates renal function in cirrhotic patients due to a number of factors: Creatinine production in patients with cirrhosis is reduced due to muscle wasting, there is an increased secretion of creatinine in the renal tubules, sCr may be diluted due to an increased volume of distribution, and finally, high bilirubin levels may interfere with the assays to measure its level. Recently, the International Club of Ascites (ICA) has adopted the concept of AKI which was developed originally to be used in general critically-ill patients. AKI is defined as the increase of at least 0.3 mg/dL (26 μmol/L) and/or ≥ 50% from baseline, within 48 hours Since urea absorption is largely modulated in the proximal tubules, it is not affected by diuretics acting more distally. The investigators therefore hypothesized that the fractional excretion of urea (FEUrea) could serve as a clinical aid in making an early distinction between ATN versus Pre renal azotemia and HRS type 1 in patients with cirrhosis and ascites presenting with AKI Fractional excretion of urea (FEUrea) ([urine urea nitrogen/ blood urea nitrogen)/(urine creatinine/plasma creatinine)] X 100) < 35% is specific for prerenal azotemia, and > 50% is specific for ATN

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis of any etiology diagnosed by clinical parameters involving laboratory tests, endoscopic or radiologic evidence of cirrhosis,
* History of decompensation (hepatic encephalopathy, ascites, variceal bleeding, jaundice)
* Age greater than 18 years
* Presence of moderate or severe ascites

Exclusion Criteria:

Patients excluded from analysis were those who did not meet inclusion criteria as well as the following

* Prior liver or kidney transplant,
* Advanced chronic kidney disease G4(GFR category grade 4) according to KDIGO guidelines.
* Patients on acute or chronic renal replacement therapy,
* Ambiguous diagnosis of AKI and phenotype of AKI,
* Patients with hepatocellular carcinoma.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: compensated and decompensated rrhotic patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
comparison of FEUrea in different types of AKI in liver cirrhosis | baseline
  measurement of FEUrea in different types of AKI in decompansated liver cirrhosis to identify its cause

REFERENCES:
- [Background] Piano S, Brocca A, Angeli P. Renal Function in Cirrhosis: A Critical Review of Available Tools. Semin Liver Dis. 2018 Aug;38(3):230-241. doi: 10.1055/s-0038-1661372. Epub 2018 Jul 24. PMID 30041275
- [Background] Durand F, Olson JC, Nadim MK. Renal dysfunction and cirrhosis. Curr Opin Crit Care. 2017 Dec;23(6):457-462. doi: 10.1097/MCC.0000000000000457. PMID 29023314
- [Background] Bucsics T, Krones E. Renal dysfunction in cirrhosis: acute kidney injury and the hepatorenal syndrome. Gastroenterol Rep (Oxf). 2017 May;5(2):127-137. doi: 10.1093/gastro/gox009. Epub 2017 Apr 24. PMID 28533910